CLINICAL TRIAL: NCT05613738
Title: Safety and Dosimetry of 177Lu-PSMA-EB-01 in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: 177Lu-PSMA-EB-01 in Patients With Metastatic Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-NM-PSMAEB01
Record Dates: First submitted 2022-10-25; First posted 2022-11-14 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Metastatic Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01 (Experimental): All patients were intravenous injected with single dose 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Interventions: Drug: 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01
- 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01 (Experimental): All patients were intravenous injected with single dose 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Interventions: Drug: 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01
- 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01 (Experimental): All patients were intravenous injected with single dose 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Interventions: Drug: 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01

INTERVENTIONS:
Drug: 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01 — All patients were intravenous injected with single dose 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Arms: 1.11 GBq (30 mCi) of 177Lu-PSMA-EB-01
Drug: 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01 — All patients were intravenous injected with single dose 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Arms: 1.85 GBq (50 mCi) of 177Lu-PSMA-EB-01
Drug: 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01 — All patients were intravenous injected with single dose 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01 then monitored at 3 hours, 24 hours, 48 hours, 72 hours, and 168 hours post-injection.
  Arms: 2.59 GBq (70 mCi) of 177Lu-PSMA-EB-01

SUMMARY:
This is a pilot study to assess the safety and measure image-based absorbed dose of 177Lu-PSMA-EB-01, a new PSMA-specific radiopharmaceutical, in patients with metastatic castration resistant prostate cancer (mCRPC) who will undergo radioligand therapy (RLT). All patients underwent 68Ga-PSMA and 18F-FDG PET/CT for selection and were randomly divided into three groups of 3 people each.The three groups received an approximately 1.11 GBq (30mCi), 1.85 GBq (50 mCi) and 2.59 GBq (70mCi) of 177Lu-PSMA-EB-01 up to 2 cycles, respectively.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent malignant tumor in men worldwide. Prostate-specific membrane antigen (PSMA), is a surface molecule specifically expressed by prostate tumors which was shown to be a valid target for radiotherapy. 177Lu-PSMA-617, a urea-based compound, provide an effective target for the treatment of metastatic castration-resistant prostate cancer. However, a major problem in the therapeutic use of 177Lu-PSMA-617 has been its short half-life and fast rate of clearance. The investigators designed and synthesized a new radiopharmaceutical, named 177Lu-PSMA-EB-01. EB（Evans Blue）can bind to albumin to slow down its plasma clearance rate, thereby increasing tumor accumulation and reducing the total dosage of Lu-177. Hence, EB-PSMA-01 may be an option for consideration due to limited supply of Lu-177, by which more patients may be benefited by this version of 177Lu-EB-PSMA-01. This study was designed to investigate the safety, dosimetry and preliminary effects of 177Lu-EB-PSMA-01 in patients with metastatic castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* progressive metastatic castration-resistant prostate cancer
* tumors with high PSMA expression confirmed on 68Ga-PSMA PET/CT

Exclusion Criteria:

* a serum creatinine level of more than 150 μmol per liter
* a hemoglobin level of less than 10.0 g/dl
* a white-cell count of less than 4.0× 109/L
* a platelet count of less than 100 × 109/L
* a total bilirubin level of more than 3 times the upper limit of the normal range
* a serum albumin level of more than 3.0 g per deciliter
* cardiac insufficiency

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Dosimetry of normal organs and tumors | through study completion, an average of 4 weeks
  The semiquantitative dosimetry will be performed based on SPECT/CT acquisitions after the first administration of 177Lu-PSMA-EB-01. The dose delivered to normal organs and tumors will be recorded.
Hematologic adverse events collection | through study completion, an average of 6 months
  Hematologic status were performed before and every 2 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0
Hepatic and renal toxic events collection | through study completion, an average of 6 months
  Liver function, and renal function were performed before and 4 weeks after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
PSA Response | through study completion, an average of 6 months
  The serum PSA response was documented semimonthly until 6 weeks after the administration of 177Lu-PSMA-EB-01. PSA response was classified as the following: partial response (PR) if PSA decrease ≥50%, progressive disease (PD) if PSA increase ≥ 25% and stable disease (SD) if PSA increase <25% or PSA decrease <50%.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zang J, Wang G, Zhao T, Liu H, Lin X, Yang Y, Shao Z, Wang C, Chen H, Chen Y, Zhu Z, Miao W, Chen X, Zhang J. A phase 1 trial to determine the maximum tolerated dose and patient-specific dosimetry of [177Lu]Lu-LNC1003 in patients with metastatic castration-resistant prostate cancer. Eur J Nucl Med Mol Imaging. 2024 Feb;51(3):871-882. doi: 10.1007/s00259-023-06470-3. Epub 2023 Oct 21. PMID 37864592